CLINICAL TRIAL: NCT01291212
Title: Efficacy of LH Activity in Low Responder Patients With Transdermal Testosterone: a Randomised Controlled Study.
Brief Title: Efficacy of Luteinizing Hormone (LH) Activity in Low Responder Patients With Transdermal Testosterone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Francisco Fábregues, Hospital Clínic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIV-01
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-01

CONDITIONS: Other Complications Associated With Artificial Fertilization
Keywords: In Vitro Fertilization; Testosterone; Ovarian Stimulation; Luteinizing Hormone
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone and FSHr (Active Comparator)
  Interventions: Drug: testosterone and FSHr alone
- testosterone and FSHr-LHr (Active Comparator)
  Interventions: Drug: Testosterone and FSHr-LHr

INTERVENTIONS:
Drug: Testosterone and FSHr-LHr — 75U of LHr added to FSHr ovarian stimulation in IVF, when testosterone was used to improve the ovarian response
  Arms: testosterone and FSHr-LHr
Drug: testosterone and FSHr alone — FSHr alone used in ovarian stimulation in IVF, when testosterone was used to improve the ovarian response
  Arms: Testosterone and FSHr

SUMMARY:
The investigators have previously demonstrated the utility of transdermal testosterone in in vitro fertilization (IVF) low responder patients. Now, the investigators want to evaluate the efficacy of luteinizing hormone (LH) activity added to recombinant follicular stimulating hormone (FSHr) during ovarian stimulation in these patients.

DETAILED DESCRIPTION:
Studies in macaques have indicated that androgens have some synergistic effects with follicular stimulating hormone (FSH) on folliculogenesis. Our previous clinical studies demonstrated the usefulness of pretreatment with transdermal testosterone in low-responder IVF patients.

There is controversy on the usefulness of recombinant luteinizing hormone (LHr) added to FSHr in ovarian stimulation of low responder patients. Thus, our present study has been designed to compare ovarian stimulation with FSHr alone versus LHr added to FSHr when transdermal testosterone pretreatment is used.

ELIGIBILITY:
Inclusion Criteria:

* Low responder patients: patients with previously canceled cycle or recovery of 3 or less oocytes

Exclusion Criteria:

* FSH > 12
* Previous ovarian surgery

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
ovarian response | within 2 weeks after begining ovarian stimulation
  number of oocytes obtained per ovarian stimulation cycle

SECONDARY OUTCOMES:
clinical pregnancy rate | within 5 weeks (plus or minus 1 week) after embryo transfer
  The number of clinical pregnancies expressed per embryo transfer cycles. Clinical pregnancy: a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy. Multiple gestational sacs are counted as one clinical pregnancy.
Implantation rate | within 5 weeks (plus/minus 1 week) after embryo transfer
  The number of gestational sacs (observed by ultrasound examination) divided by the number of embryos transferred.
Live birth rate | within 9 months (plus/minus 1 month) after embryo transfer
  The number of deliveries that resulted in at least one live born baby expressed per 100 embryo transfer cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Balasch J, Fabregues F, Penarrubia J, Carmona F, Casamitjana R, Creus M, Manau D, Casals G, Vanrell JA. Pretreatment with transdermal testosterone may improve ovarian response to gonadotrophins in poor-responder IVF patients with normal basal concentrations of FSH. Hum Reprod. 2006 Jul;21(7):1884-93. doi: 10.1093/humrep/del052. Epub 2006 Mar 3. PMID 16517559
- [Result] Fabregues F, Penarrubia J, Creus M, Manau D, Casals G, Carmona F, Balasch J. Transdermal testosterone may improve ovarian response to gonadotrophins in low-responder IVF patients: a randomized, clinical trial. Hum Reprod. 2009 Feb;24(2):349-59. doi: 10.1093/humrep/den428. Epub 2008 Dec 3. PMID 19054777